CLINICAL TRIAL: NCT02451839
Title: An ObserVatIonal STudy of the Effectiveness of AdaLimumab on Health and Disability Outcomes in New Zealand Patients With Immune-Mediated InflammaTorY Diseases (VITALITY)
Acronym: VITALITY
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-345
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2018-01

CONDITIONS: Crohn's Disease; Rheumatoid Arthritis; Psoriasis
Keywords: Crohn Disease; Arthritis, Rheumatoid; Psoriasis; Patient Outcome Assessment; Adalimumab; Global Health; Quality of Life
MeSH Terms: conditions — Crohn Disease; Arthritis, Rheumatoid; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Crohn's Disease: Participants with Crohn's disease. All participants will receive at least 3 months of treatment with adalimumab. Adalimumab was prescribed by the physician under usual and customary practice and according to the approved adalimumab New Zealand Datasheet.
- Rheumatoid Arthritis: Participants with rheumatoid arthritis. All participants will receive at least 3 months of treatment with adalimumab. Adalimumab was prescribed by the physician under usual and customary practice and according to the approved adalimumab New Zealand Datasheet.
- Psoriasis: Participants with psoriasis. All participants will receive at least 3 months of treatment with adalimumab. Adalimumab was prescribed by the physician under usual and customary practice and according to the approved adalimumab New Zealand Datasheet.

SUMMARY:
For public health purposes disability is becoming increasingly important as an outcome measure. Despite this, there are few data on the effectiveness of adalimumab on disability outcomes in patients with immune-mediated inflammatory diseases (IMIDs), particularly in the Phase IV setting. There are even less data available in New Zealand, which did not have the opportunity to participate to a major extent in large, multinational, Phase III pivotal studies of adalimumab in IMIDs.

The World Health Organisation Disability Assessment Schedule (WHODAS) 2.0 is a simple, validated, free and easy-to-use generic assessment instrument for health and disability. It is applicable across cultures, in all adult populations. It is a responsive measure that can show what difference a treatment makes.

Results from study of effect of adalimumab on WHODAS scores and other patient-reported outcomes (PROs) of work activity and well-being will be of interest to a variety of stakeholders in the healthcare system including patients, healthcare practitioners and payers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of rheumatoid arthritis, Crohn's disease or psoriasis who have made a decision with their physician to commence treatment with adalimumab in accordance with routine medical practice and with the approved adalimumab New Zealand Datasheet.
* Patients who have been evaluated for tuberculosis risk factors/exposure for active/latent tuberculosis infection (per local requirements and according to the approved adalimumab New Zealand Datasheet).
* Adult subjects, 18-75 years old, who have voluntarily signed and dated an informed consent form prior to any study-specific procedures.

Exclusion Criteria:

* Previous treatment with adalimumab.
* Previous treatment with any biologic.
* Severe infection including sepsis, active tuberculosis or opportunistic infection.
* Moderate to severe heart failure (New York Heart Association Class II/III).
* Concurrent administration with anakinra.
* Hypersensitivity to adalimumab or its excipients.
* Any condition that in the opinion of the investigator would compromise the subject's well-being or ability to perform the study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be males and/or females who are attending a routine clinical visit and meet all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gearry RB, Frampton C, Inns S, Poppelwell D, Rademaker M, Suppiah R. VITALITY: impact of adalimumab on health and disability outcomes in patients with Crohn's disease, rheumatoid arthritis, or psoriasis treated in clinical practice in New Zealand. Curr Med Res Opin. 2019 Oct;35(10):1837-1846. doi: 10.1080/03007995.2019.1634952. Epub 2019 Jul 3. PMID 31233347
- See also: http://rxabbvie.com/ — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 168 recruited participants, 4 withdrew or were withdrawn prior to baseline measures being completed (164 participants had baseline World Health Organization Disability Assessment Schedule [WHODAS] data recorded).
Groups:
- Crohn's Disease: Participants with Crohn's disease. All participants received at least 3 months of treatment with adalimumab. Adalimumab was prescribed by the physician under usual and customary practice and according to the approved adalimumab New Zealand Datasheet.
- Rheumatoid Arthritis: Participants with rheumatoid arthritis. All participants received at least 3 months of treatment with adalimumab. Adalimumab was prescribed by the physician under usual and customary practice and according to the approved adalimumab New Zealand Datasheet.
- Psoriasis: Participants with psoriasis. All participants received at least 3 months of treatment with adalimumab. Adalimumab was prescribed by the physician under usual and customary practice and according to the approved adalimumab New Zealand Datasheet.
Period: Overall Study
Arm/Group | Crohn's Disease | Rheumatoid Arthritis | Psoriasis
Started | 72 | 59 | 37
Baseline WHODAS Data Recorded | 70 | 57 | 37
Completed | 44 | 40 | 30
Not Completed | 28 | 19 | 7

BASELINE CHARACTERISTICS:
Population: Participants with baseline WHODAS data recorded. Per protocol, primary and secondary endpoint data [other than the endpoints presented in Outcome Measures 4-6 and 14-16] were intended to be analyzed across all indications; therefore, corresponding baseline data are presented for all participants as a single group.
Groups:
- All Indications: Participants with Crohn's disease, rheumatoid arthritis, or psoriasis. All participants received at least 3 months of treatment with adalimumab. Adalimumab was prescribed by the physician under usual and customary practice and according to the approved adalimumab New Zealand Datasheet.
Arm/Group | All Indications
Number analyzed (Participants) | 164
Age, Continuous [Mean (Full Range); unit: years] | 45.7 [16.9 to 77.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5
  European | 145
  Maori | 7
  Other (Not Specified) | 4
  Pacific Peoples | 3
World Health Organization Disability Assessment Schedule (WHODAS) 2.0 Response Score [Mean (Standard Deviation); unit: units on a scale] — WHODAS 2.0 is a measures health and disability across cultures in all adult populations by assessing the same individual before and after the intervention across 12 items, covering the following 6 domains: cognition, mobility, self-care, getting along, life activities and participation. Scores assigned to each of the items (none=0, mild=1, moderate=2, severe=3, and extreme=4) are summed. Scores can range from 0 to 48. Persons scoring 10 to 48 are likely to have clinically significant disability. Population: Participants with baseline and Month 6 assessments in each of the indication categories.
  units on a scale
    All Indications: number analyzed (Participants) | 114
    All Indications | 15.2 (9.1)
    Crohn's disease: number analyzed (Participants) | 44
    Crohn's disease | 13.2 (7.3)
    Rheumatoid arthritis: number analyzed (Participants) | 40
    Rheumatoid arthritis | 17.9 (8.1)
    Psoriasis: number analyzed (Participants) | 30
    Psoriasis | 14.4 (11.7)
Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH) V2.0: Absenteeism [Mean (Standard Deviation); unit: percentage of work time missed] — WPAI:GH is a 6-item questionnaire looks at the effect of health problems on ability to work and perform regular activities. The WPAI yields 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. The questionnaire specifies responses for the previous 7 days. Population: Participants with a baseline and Month 6 assessment.
  percentage of work time missed
    number analyzed (Participants) | 68
    (all) | 14.7 (30.0)
WPAI-GH v2.0: Presenteeism [Mean (Standard Deviation); unit: percentage impairment time] — WPAI:GH is a 6-item questionnaire looks at the effect of health problems on ability to work and perform regular activities. The WPAI yields 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. The questionnaire specifies responses for the previous 7 days. Population: Participants with a baseline and Month 6 assessment.
  percentage impairment time
    number analyzed (Participants) | 71
    (all) | 39.7 (28.8)
WPAI-GH v2.0: Work Productivity Loss [Mean (Standard Deviation); unit: percentage overall work impairment] — WPAI:GH is a 6-item questionnaire looks at the effect of health problems on ability to work and perform regular activities. The WPAI yields 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. The questionnaire specifies responses for the previous 7 days. Population: Participants with a baseline and Month 6 assessment.
  percentage overall work impairment
    number analyzed (Participants) | 68
    (all) | 29.4 (22.5)
WPAI-GH v2.0: Activity Impairment [Mean (Standard Deviation); unit: percentage of activity impairment] — WPAI:GH is a 6-item questionnaire looks at the effect of health problems on ability to work and perform regular activities. The WPAI yields 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. The questionnaire specifies responses for the previous 7 days. Population: Participants with a baseline and Month 6 assessment.
  percentage of activity impairment
    number analyzed (Participants) | 114
    (all) | 51.9 (28.1)
Kessler Psychological Distress Scale (K10) [Mean (Standard Deviation); unit: units on a scale] — The K10 questionnaire is intended to yield a global measure of distress based on questions about anxiety and depressive symptoms that a person has experienced in the most recent 4-week period. In this 10-item questionnaire, scores are summed and range from 10 to 50. Patients with a score under 20 are likely to be well, those with a score 20-24 are likely to have a mild mental disorder, those with a score 25-29 are likely to have a moderate mental disorder and those with a score 30 and over are likely to have a severe mental disorder. Population: Participants with a baseline and Month 6 assessment.
  units on a scale
    number analyzed (Participants) | 114
    (all) | 23.0 (8.2)
Flourishing Scale [Mean (Standard Deviation); unit: units on a scale] — The Flourishing Scale consists of eight items describing important aspects of human functioning ranging from positive relationships, to feelings of competence, to having meaning and purpose in life. Patients respond to the eight questions using responses varying between 1 (strongly disagree) and 7 (strongly agree). For the scoring, the responses are added such that the range of scores is 8 (lowest possible) to 56 (highest possible). While there is no set cut point to define disability, a high score represents a person with many psychological resources and strengths. Population: Participants with a baseline and Month 6 assessment.
  units on a scale
    number analyzed (Participants) | 114
    (all) | 45.0 (9.0)
Subjective Vitality Scale [Mean (Standard Deviation); unit: units on a scale] — The Subjective Vitality Scale assesses the state of feeling alive and alert to having energy available to the self. Patients respond to eight prompts, with a response ranging from 1=strongly disagree to 7=strongly agree. The sum of the scores is calculated with a higher score indicating a better condition. Population: Participants with a baseline and Month 6 assessment.
  units on a scale
    number analyzed (Participants) | 113
    (all) | 25.4 (7.4)
Health Assessment Questionnaire Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — HAQ-DI measures functional status in rheumatic diseases. It has 20 items, and asks patients to report the degree of difficulty faced in several areas of their life including: dressing and grooming, arising, eating, walking, hygiene, reach, grip, activities based on the previous week on a scale from 0 (without any difficulty) to 3 (cannot be done at all). It also asks the participant to rate their pain and health in the previous week. Scores on each task are summed and averaged to provide an overall score ranging from 0 (no disability) to 3 (very severe, high-dependency disability). Population: Participants with rheumatoid arthritis and a baseline and Month 6 assessment.
  units on a scale
    number analyzed (Participants) | 40
    (all) | 1.9 (0.6)
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) [Mean (Standard Deviation); unit: units on a scale] — The SIBDQ is a simple validated, 10-item questionnaire designed to find out how the patient has been feeling in the previous 2 weeks. Quality of life (QoL) is measured in 4 domains: bowel symptoms, emotional health, systemic systems and social function. Participants respond to questions ranging from 1=all of the time to 7=none of the time. Scores are added together, with higher scores indicating a better health-related QoL. Total scores range from 10 (poor QoL) to 70 (good QoL). Population: Participants with Crohn's disease and baseline and Month 6 assessments.
  units on a scale
    number analyzed (Participants) | 43
    (all) | 36.1 (9.7)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: units on a scale] — The DLQI measures 10 items covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, to determine how much the patients skin problem affected their life in the past week. Participants respond to the questions with 'very much,' 'a lot,' 'a little,' or 'not at all.' The scores are added together, and the impact on QoL is banded as follows: 0-1=no effect on participant's life; 2-5=small effect; 6-10=moderate effect; 11-20=very large effect; 21-30=extremely large effect. Population: Participants with psoriasis and a baseline and Month 6 assessment.
  units on a scale
    number analyzed (Participants) | 30
    (all) | 15.8 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WHODAS 2.0 Response Score at Month 6 Across All Indications
Description: WHODAS 2.0 is a measures health and disability across cultures in all adult populations by assessing the same individual before and after the intervention across 12 items, covering the following 6 domains: cognition, mobility, self-care, getting along, life activities and participation. Scores assigned to each of the items (none=0, mild=1, moderate=2, severe=3, and extreme=4) are summed. Scores can range from 0 to 48. Persons scoring 10 to 48 are likely to have clinically significant disability.
Time Frame: Baseline, Month 6
Population: Participants with baseline and Month 6 assessments. Per protocol, primary and secondary endpoint data [other than the endpoints presented in Outcome Measures 4-6 and 14-16] were intended to be analyzed across all indications; therefore, data are presented for all participants as a single group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Indications
Number analyzed (Participants) | 114
units on a scale | 7.9 (8.1)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p < 0.001, paired t-test

2. Secondary Outcome: Change From Baseline in WHODAS 2.0 Response Score at Month 2 Across All Indications
Description: as for outcome 1
Time Frame: Baseline, Month 2
Population: Participants with baseline and Month 2 assessments. Per protocol, primary and secondary endpoint data [other than the endpoints presented in Outcome Measures 4-6 and 14-16] were intended to be analyzed across all indications; therefore, data are presented for all participants as a single group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Indications
Number analyzed (Participants) | 130
units on a scale | 5.7 (8.0)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p < 0.001, paired t-test

3. Secondary Outcome: Change From Baseline in WHODAS 2.0 Response Score at Month 4 Across All Indications
Description: as for outcome 1
Time Frame: Baseline, Month 4
Population: Participants with baseline and Month 4 assessments. Per protocol, primary and secondary endpoint data [other than the endpoints presented in Outcome Measures 4-6 and 14-16] were intended to be analyzed across all indications; therefore, data are presented for all participants as a single group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Indications
Number analyzed (Participants) | 115
units on a scale | 7.1 (8.4)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p < 0.001, paired t-test

4. Secondary Outcome: Change From Baseline in WHODAS 2.0 Response Score at Month 6 in Participants With Crohn's Disease
Description: as for outcome 1
Time Frame: Baseline, Month 6
Population: Participants with Crohn's disease and baseline and Month 6 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 44
units on a scale | 6.3 (7.3)
Statistical Analysis 1: Comparison: Crohn's Disease; Test type: Superiority; p < 0.001, paired t-test

5. Secondary Outcome: Change From Baseline in WHODAS 2.0 Response Score at Month 6 In Participants With Psoriasis
Description: as for outcome 1
Time Frame: Baseline, Month 6
Population: Participants with psoriasis and baseline and Month 6 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoriasis
Number analyzed (Participants) | 30
units on a scale | 8.1 (8.9)
Statistical Analysis 1: Comparison: Psoriasis; Test type: Superiority; p < 0.001, paired t-test

6. Secondary Outcome: Change From Baseline in WHODAS 2.0 Response Score at Month 6 in Participants With Rheumatoid Arthritis
Description: as for outcome 1
Time Frame: Baseline, Month 6
Population: Participants with rheumatoid arthritis and baseline and Month 6 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 40
units on a scale | 9.5 (8.3)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis; Test type: Superiority; p < 0.001, paired t-test

7. Secondary Outcome: Change From Baseline in WPAI:GH V2.0 Score at Month 6 Across All Indications: Absenteeism
Description: WPAI:GH is a 6-item questionnaire looks at the effect of health problems on ability to work and perform regular activities. The WPAI yields 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. The questionnaire specifies responses for the previous 7 days.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | All Indications
Number analyzed (Participants) | 68
percentage of work time missed | 10.6 (34.7)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p = 0.015, paired t-test

8. Secondary Outcome: Change From Baseline in WPAI:GH V2.0 Score at Month 6 Across All Indications: Presenteeism
Description: as for outcome 7
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage impairment time
Arm/Group | All Indications
Number analyzed (Participants) | 71
percentage impairment time | 18.0 (33.1)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p < 0.001, paired t-test

9. Secondary Outcome: Change From Baseline in WPAI:GH 2.0 Score at Month 6 Across All Indications: Work Productivity Loss
Description: as for outcome 7
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage overall work impairment
Arm/Group | All Indications
Number analyzed (Participants) | 68
percentage overall work impairment | 9.7 (28.0)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p = 0.006, paired t-test

10. Secondary Outcome: Change From Baseline in WPAI:GH V2.0 Score at Month 6 Across All Indications: Activity Impairment
Description: as for outcome 7
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of activity impariment
Arm/Group | All Indications
Number analyzed (Participants) | 114
percentage of activity impariment | 24.1 (34.0)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p < 0.001, paired t-test

11. Secondary Outcome: Change From Baseline in K10 at Month 6 Across All Indications
Description: The K10 is intended to yield a global measure of distress based on a questionnaire about anxiety and depressive symptoms that a person has experienced in the most recent 4 week period. The K10 scale involves 10 questions about emotional states each with a 5-level response scale. Each item is scored from 1=none of the time to 5=all of the time. Scores of the 10 items are then summed, yielding a minimum score of 10 and a maximum score of 50. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Indications
Number analyzed (Participants) | 114
units on a scale | 6.1 (7.7)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p < 0.001, paired t-test

12. Secondary Outcome: Change From Baseline in Flourishing Scale at Month 6 Across All Indications
Description: The Flourishing Scale is a brief 8-item summary measure of the respondent's self-perceived success in important areas such as relationships, self-esteem, purpose, and optimism. The scale provides a single psychological well-being score. Participants are asked to respond to 8 statements using a scale of 1 (strongly disagree) and 7 (strongly agree) for each item. The possible range of scores is from 8 (lowest possible) to 56 (highest possible), with higher scores representing more psychological resources and strengths.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Indications
Number analyzed (Participants) | 114
units on a scale | -2.3 (8.7)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p = 0.006, paired t-test

13. Secondary Outcome: Change From Baseline in Subjective Vitality Scale at Month 6 Across All Indications
Description: The Subjective Vitality Scale assesses the state of feeling alive and alert to having energy available to the self. Patients respond to eight prompts, with a response ranging from 1=strongly disagree to 7=strongly agree. The sum of the scores is calculated with a higher score indicating a better condition. The total score ranges from 8 to 56 with a higher score indicating a better condition.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Indications
Number analyzed (Participants) | 113
units on a scale | -5.4 (8.3)
Statistical Analysis 1: Comparison: All Indications; Test type: Superiority; p < 0.001, paired t-test

14. Secondary Outcome: Change From Baseline in HAQ-DI Score at Month 6 in Participants With Rheumatoid Arthritis
Description: HAQ-DI measures functional status in rheumatic diseases. It has 20 items, and asks patients to report the degree of difficulty faced in several areas of their life including: dressing and grooming, arising, eating, walking, hygiene, reach, grip, activities based on the previous week on a scale from 0 (without any difficulty) to 3 (cannot be done at all). It also asks the participant to rate their pain and health in the previous week. Scores on each task are summed and averaged to provide an overall score ranging from 0 (no disability) to 3 (very severe, high-dependency disability).
Time Frame: Baseline, Month 6
Population: Participants with rheumatoid arthritis baseline and Month 6 assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 40
score on a scale | 0.4 (0.4)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis; Test type: Superiority; p < 0.001, paired t-test

15. Secondary Outcome: Change From Baseline in SIBDQ Score at Month 6 in Participants With Crohn's Disease
Description: The SIBDQ is a simple validated, 10-item questionnaire designed to find out how the patient has been feeling in the previous 2 weeks. QoL is measured in 4 domains: bowel symptoms, emotional health, systemic systems and social function. Participants respond to questions ranging from 1=all of the time to 7=none of the time. Scores are added together, with higher scores indicating a better health-related QoL. Total scores range from 10 (poor QoL) to 70 (good QoL).
Time Frame: Baseline, Month 6
Population: Participants with Crohn's disease and baseline and Month 6 assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 43
score on a scale | -16.3 (13.7)
Statistical Analysis 1: Comparison: Crohn's Disease; Test type: Superiority; p < 0.001, paired t-test

16. Secondary Outcome: Change From Baseline in DLQI Score at Month 6 in Participants With Psoriasis
Description: The DLQI measures 10 items covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, to determine how much the patients skin problem affected their life in the past week. Participants respond to the questions with 'very much,' 'a lot,' 'a little,' or 'not at all.' The scores are added together, and the impact on QoL is banded as follows: 0-1=no effect on participant's life; 2-5=small effect; 6-10=moderate effect; 11-20=very large effect; 21-30=extremely large effect.
Time Frame: Baseline, Month 6
Population: Participants with psoriasis and baseline and Month 6 assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriasis
Number analyzed (Participants) | 30
score on a scale | 11.0 (7.6)
Statistical Analysis 1: Comparison: Psoriasis; Test type: Superiority; p < 0.001, paired t-test

17. Secondary Outcome: Number of Participants Remaining on Treatment at Month 6
Description: The number of participants at 6 months who remained on adalimumab, having satisfied the requirements for application for renewal of subsidy by special authority.
Time Frame: Month 6
Population: Participants completing the study at 6 months. Per protocol, primary and secondary endpoint data [other than the endpoints presented in Outcome Measures 4-6 and 14-16] were intended to be analyzed across all indications; therefore, data are presented for all participants as a single group.
Measure: Count of Participants; unit: Participants
Arm/Group | All Indications
Number analyzed (Participants) | 114
Participants | 108

ADVERSE EVENTS:
Time Frame: From the signing of informed consent through Month 6
Description: Per protocol, adverse event data were intended to be analyzed across all indications; therefore, data are presented for all participants as a single group.
Arm/Group | All Indications
All-Cause Mortality (participants affected / at risk) | 1/164
Serious Adverse Events (participants affected / at risk) | 18/164
Other Adverse Events (participants affected / at risk) | 65/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Indications (N=164)
Crohn's disease (Gastrointestinal disorders) | 3
Gastritis erosive (Gastrointestinal disorders) | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1
Ileal stenosis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Abdominal hernia (General disorders) | 1
Death (General disorders) | 1 — death due to unknown cause
Non-cardiac chest pain (General disorders) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Stoma complication (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Indications (N=164)
Angina pectoris (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Eye irritation (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Aphthous ulcer (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Drug intolerance (General disorders) | 1
Fatigue (General disorders) | 3
Influenza like illness (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site reaction (General disorders) | 4
Injection site urticaria (General disorders) | 2
Malaise (General disorders) | 1
Pain (General disorders) | 3
Ulcer (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Adenovirus infection (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Kidney infection (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis streptococcal (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Tinea pedis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Glycosylated haemoglobin increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Peyronie's disease (Reproductive system and breast disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT02451839/Prot_SAP_000.pdf